CLINICAL TRIAL: NCT05800496
Title: A Proof-of-Concept, Placebo-Controlled, Safety, and Efficacy Study of Plant Based Biotin in Healthy Adult Human Subjects With Thin, Dry, and Brittle Hair
Brief Title: A Clinical Study to Assess the Safety and Effectiveness of Plant Based Biotin in Healthy Human Subjects With Thin, Dry, and Brittle Hair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: ZYWIE VENTURES PRIVATE LIMITED (Unknown)
Responsible Party: Principal Investigator, Dr Nayan Patel, Principal Investigator-Medical Director, NovoBliss Research Pvt Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NB220024-FC
Record Dates: First submitted 2023-02-25; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Hair Thinning; Hair Brittle; Dry Hair
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: A Proof-of-Concept, Placebo-Controlled, Safety, and Efficacy
Who Masked: Participant, Investigator
Masking Description: Subjects were randomly assigned in a 1:1 ratio to receive either treatment A or Placebo. The randomization code was generated by NovoBliss Research.
  Subjects were randomly allocated to one of the treatment groups, as per the randomization code. Complete double-blinding was kept wherein neither the subjects nor the investigator was aware of the test treatment allocation. To maintain double blinding, the study staff who involves in treatment dispensing and distribution was not involved in any other study-related activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SesZen-Bio™ (Experimental): SesZen-Bio™ is specially formulated for healthy hairs and healthy skin. Fortified with Sesbania Agati for 2X Hair Follicle Stimulation & Hair Fall Control, to Promote Shiny Hair, biotin that Supports Hair Growth.
  Interventions: Dietary Supplement: SesZen-Bio™
- Placebo (Tapioca based starch Capsules) (Placebo Comparator): tapioca starch, is a starchy white flour that has a slight sweet flavor to it and is prepared by extrusion and coating process.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: SesZen-Bio™ — mode of usage: 1 capsule in the morning and 1 capsule at night. administration: Oral Administration
  Arms: SesZen-Bio™
Other: Placebo — Mode of Usage: 1 capsule in the morning and 1 capsule at night. Route of Administration: Oral Administration
  Arms: Placebo (Tapioca based starch Capsules)

SUMMARY:
This is a randomized, placebo-controlled, double-blind, two-arm, single-centre, proof-of-concept, clinical study to evaluate the safety and efficacy of Plant based Biotin in Healthy Human Subjects with thin, dry, and brittle hair.

a sufficient number (maximum of 54 (27/arm)) of female/male adult subjects were recruited/enrolled to ensure a total of 50 subjects (25 subjects/arm) completed the study.

DETAILED DESCRIPTION:
This is a randomised, placebo-controlled, double-blind, two-arm, single-centre, proof-of-concept, clinical study to evaluate the safety and efficacy of Plant based Biotin in Healthy Human Subjects with thin, dry and brittle hair.

a sufficient number (maximum of 54 (27/arm)) of female/male adult subjects were recruited/enrolled to ensure a total of 50 subjects (25 subjects/arm) completed the study.

total of 51 subjects was completed the study. The potential subjects were screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. The adult female/male subjects were instructed to visit the facility as per the below visits.

* Visit 01 (Day 01): Screening, Enrolment, Baseline Evaluations
* Visit 02 (Day 28): Treatment Period, Evaluations
* Visit 03 (Day 56): Evaluations, End of Study Visit Subjects were pre-screened by the screening department of NovoBliss Research. Subjects were called on the telephone by the recruiting department prior to the enrolment visit. Subjects were told during screening (prior to enrolment) not to wear any facial make-up or use any hair product on the study visit day.

Assessment of efficacy parameters before test treatment usage was done on day 1, and after test treatment usage was done on day 28, and day 56 as listed below.

* General Appearance of Hair i.e., hair volume, hair reflection, hair plasticity, hair density, hair smoothness, hair oiliness, hair shininess.
* General Appearance of Scalp i.e., Scalp itchiness, redness, scaling.
* CASLite Nova: Hair Density, Thickness, scalp condition
* Visioscan (C+K Instrument): Crow's feet area wrinkles, fine lines, skin texture - roughness,
* Skin Colorimeter CL 400: Right cheek skin colour evenness L*, a* b* and RGB, ITA Angle
* DermaLab®Combo - skin elasticity (Right cheek)
* MoitureMeterEPiD: Skin Hydration (Right cheek)
* Vapometer: Skin Barrier function - Transepidermal water loss (Right cheek)
* Physician Global Assessment for improvement in brittle nails - Day 01 and Day 56
* Serum Ferratin Biomarker test (Day 1 as baseline and Day 56)
* Digital Photographs: Facial photographs Before test treatment usage and after test treatment usage.
* Subjective Product Perception Assessment regarding the test product's effect on hair and skin firmness, appearance, nails etc

ELIGIBILITY:
Inclusion Criteria:

1. Age: 30 to 55 years (both inclusive) at the time of consent.
2. Sex: Healthy males and non-pregnant/non-lactating females.
3. Females of childbearing potential must have a self-reported negative pregnancy test.
4. Subjects are generally in good health.
5. Subject with self-proclaimed nonpathological thin, dry and brittle hair.
6. Subject with normal Fitzpatrick skin type III to VI (Human skin colour determination scale).
7. Subject has a score of at least "mild skin aging" based on PGA at screening visit.
8. Subject with Glogau Skin Age II or III as assessed by the Dermatologist/ Dermatologist Trained Evaluator.
9. Subject is willing to forgo cosmetic procedures 3 months prior to and for the duration of the study.
10. Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
11. Subject is able to follow their normal skin care routines and to refrain from introducing any new skin care products during the study.
12. Subject is able to forgo changes in baseline medications and nutritional supplements during the study period.
13. If the subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post- menopausal for at least 1 year or have had a tubal ligation.
14. If currently using hormonal contraception, has been using this form of contraception for at least 6 months and agrees to continue using the same contraception for the duration of the study.
15. Subjects are willing not to introduce any new soaps, cleansers, laundry detergents, lotions, creams, shampoos etc. for the duration of the study.
16. Subjects are willing to give written informed consent and are willing to follow the study procedure.
17. Subjects who have used other marketed products for hair thinning in the past.
18. Subjects who commit not to use medicated/ prescription shampoos/hair care products (containing Minoxidil / Anti-thinning agents) or any other hair growth, treatment for thin hair, or hair products other than the test product for the entire duration of the study.
19. Willing to use test product throughout the study period

Exclusion Criteria:

1. Subjects with a history of hair thinning/hair fall due to any clinically significant problems/s like anaemia, thyroid problems, etc.
2. Subject has a history of allergy or sensitivity to the test treatment ingredients like sesbania agati and others etc.
3. Subject has a history of any dermatological condition of the scalp other than hair loss and/or dandruff or active dermatological condition that might interfere with the clinical assessments (e.g. tattoos, eczema, psoriasis, acne, etc.).
4. Subject has used any systemic therapy with chronic antibiotic therapy, retinoids, and/or oral steroids during the 4 weeks prior to the start or anticipates having to use at any point during the study.
5. Subject has applied any topical retinoids within 2 weeks of the screening visit or anticipates having to use at any point during the study.
6. Subject is not willing to avoid unprotected sun or other UV radiation exposure during the study period.
7. Subject is currently pregnant/breastfeeding.
8. Subject has a history of prior use of hair growth treatment within 3 months.
9. Subject has a history of any prior hair growth procedures (e.g., hair transplant or laser).
10. Subject has a history of alcohol or drug addiction.
11. Subjects who have plans of shaving scalp hair during the study.
12. Subject has a past or present condition of irritated or visibly inflamed scalp or severe scalp disease.
13. Subject who is currently participating in or planning on starting weight loss program that may result in a significant change in overall body weight.
14. Any other condition which could warrant exclusion from the study, as per the dermatologist's/investigator's discretion.
15. Pregnant or breastfeeding or planning to become pregnant during the study period.
16. History of chronic illness which may influence the cutaneous state.
17. Subjects participating in other similar cosmetics, devices or therapeutic trials or hair/scalp/skin care products within the last four weeks.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Change in Hair Density | Day 01,Day 28 (+ 02 Days) and Day 56 (+ 02 Days)
  To evaluate the effectiveness of test treatment in terms of change in hair density between the treatment and placebo group by using CasaLiteNova (Instrumental Reading)
Change in Hair Thickness | Day 01, Day 28 (+ 02 Days) and Day 56 (+ 02 Days)
  To evaluate the effectiveness of test treatment in terms of change in hair thickness between the treatment and placebo group by using CasaLiteNova (Instrumental Reading)
Change in Scalp Condition | Day 01, Day 28 (+ 02 Days) and Day 56 (+ 02 Days)
  To evaluate the effectiveness of test treatment in terms of change in scalp condition between the treatment and placebo group by using CasaLiteNova (Instrumental Reading)
Change in Facial Wrinkle | Day 01, Day 28 (+ 02 Days) and Day 56 (+ 02 Days)
  To evaluate the effectiveness of test treatment in terms of reducing facial wrinkle between the treatment and placebo group by using VisioScan (Instrumental Readings)
Change in Fine Lines | Day 01, Day 28 (+ 02 Days) and Day 56 (+ 02 Days)
  To evaluate the effectiveness of test treatment in terms of reducing fine lines between the treatment and placebo group by using VisioScan (Instrumental Readings)

SECONDARY OUTCOMES:
Change in Physician Global Assessment (PGA) scoring | Day 01, Day 28 (+ 02 Days) and Day 56 (+ 02 Days)
  To assess the effectiveness of test treatment in terms of change in Physician Global Assessment (PGA) between the treatment and placebo group by using Griffiths Scale 0 point= No appearance, 7-9point= Severe
Change in Glogau Skin Age | Day 01, Day 28 (+ 02 Days) and Day 56 (+ 02 Days)
  To assess the effectiveness of test treatment in terms of change in Glogau Skin Age between the treatment and placebo group by using Glogau Skin Age Classification
Change in Skin Colour | Day 01, Day 28 (+ 02 Days) and Day 56 (+ 02 Days)
  To assess the effectiveness of test treatment in terms of change in skin colour between the treatment and placebo group i.e.L* a* b* and ITA (Individual Topology Angle) using Skin-Colorimeter CL 400 (Instrumental Readings)
Change in Skin Elasticity | Day 01, Day 28 (+ 02 Days) and Day 56 (+ 02 Days)
  To assess the effectiveness of test treatment in terms of change in skin elasticity between the treatment and placebo group by using DermaLab Combo (Instrumental Reading)
Change in Skin Hydration | Day 01, Day 28 (+ 02 Days) and Day 56 (+ 02 Days)
  To assess the effectiveness of test treatment in terms of change in skin hydration between the treatment and placebo group by using MoistureMeterEpiD (Instrumental Reading) the result indicated in %
Change in Skin barrier Function | Day 01, Day 28 (+ 02 Days) and Day 56 (+ 02 Days)
  To assess the effectiveness of test treatment in terms of change in Skin Barrier Function between the treatment and placebo group by using Vapometer (Instrumental Reading) the result indicated in %
Change in Serum Ferritin | Day 01, Day 28 (+ 02 Days) and Day 56 (+ 02 Days)
  To assess the effectiveness of test treatment in terms of change in serum ferritin between the treatment and placebo group
Change in brittle nails | Day 01, Day 28 (+ 02 Days) and Day 56 (+ 02 Days)
  To assess the effectiveness of test treatment in terms of change in brittle nails between the treatment and placebo group by using Physician Global Assessment (PGA) 0=None, 5= Severe
Noticeable Improvement in Facial Photograph | Day 01, Day 28 (+ 02 Days) and Day 56 (+ 02 Days)
  To assess the effectiveness of test treatment in terms of noticeable improvement in Facial Wrinkle between the treatment and placebo group by using Digital Camera (Visual Change)
Subjective Perception Questionnaires | Day 01, Day 28 (+ 02 Days) and Day 56 (+ 02 Days)
  To assess the effectiveness of test treatment in terms of Subjective perception on color, fragrance, taste, skin hydration, skin tone, firmness, appearance, hair and nails strongness and shine between the treatment and placebo group by using 9 point Hedonic scale

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Nayan K Patel, MBBS, Principal Investigator — Medical Director
Locations (1):
- NovoBliss Research Pvt Ltd, Gandhinagar, Gujarat, India

IPD SHARING:
Plan to Share IPD: No